CLINICAL TRIAL: NCT06081413
Title: Bariatric and Metabolic Surgery in Patients Over 65 Years of Age - a Multicenter Study
Brief Title: Bariatric and Metabolic Surgery in Patients Over 65 Years of Age
Acronym: 65plus
Status: Completed | Type: Observational
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Responsible Party: Principal Investigator, Natalia Dowgiałło-Gornowicz, MD, PhD, assistant professor, University of Warmia and Mazury in Olsztyn
Other Study IDs: 38/2023
Record Dates: First submitted 2023-10-02; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Hypertension
Keywords: bariatric surgery; elderly patients; obesity-related diseases
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Hypertension | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric surgery — bariatric surgeries - sleeve gastrectomy, roux-en-Y gastric bypass, one anastomosis gastric bypass, adjustable gastric band

SUMMARY:
A retrospective multicenter study that will analyze the results of surgical treatment of obesity in patients over 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and more
* undergone bariatric surgery

Exclusion Criteria:

* lost to follow up

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: all patients over 65 years of age who underwent bariatric procedures
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
weight loss after bariatric surgery | until December 31, 2022
  how much weight patients lost, determined by BMI
improvement in obesity-related diseases | until December 31, 2022
  changes in the treatment of hypertension and diabetes type 2 - whether the diseases resolved completely or whether there was a change in medications (in accordance with the guidelines of the American Society for Metabolic and Bariatric Surgery ASMBS)

CONTACTS AND LOCATIONS:
Locations (1):
- UWM, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: No